CLINICAL TRIAL: NCT00154830
Title: Alterations of Functional Activities and Leg Stiffness After Hamstring Lengthening in Cerebral Palsy Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9200201507
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-11-23 (Estimated); Status verified 2005-07

CONDITIONS: Cerebral Palsy; Crouch Gait
MeSH Terms: conditions — Cerebral Palsy

INTERVENTIONS:
Behavioral: cerebral palsy
Behavioral: crouch gait

SUMMARY:
Cerebral palsy (CP) is the most prevalent physical disabilities originating in childhood. Crouch gait is a common gait abnormality in patients with cerebral palsy, which is common treated with hamstring lengthening. This surgery can alter mechanical property of lower limb and affected ability of generating force in hamstring, leading changes in functional activities. Therefore, the first aim of this study is to investigate the effects of hamstring lengthening on pelvis and hip control while performing functional activity, including level walking and sit-to-stand.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most prevalent physical disabilities originating in childhood. Crouch gait is a common gait abnormality in patients with cerebral palsy, which is common treated with hamstring lengthening. This surgery can alter mechanical property of lower limb and affected ability of generating force in hamstring, leading changes in functional activities. Therefore, the first aim of this study is to investigate the effects of hamstring lengthening on pelvis and hip control while performing functional activity, including level walking and sit-to-stand.

Gait or motion analysis has been used widely in the diagnosis of patients with locomotor pathology and the subsequent planning and assessment of treatment. Ten subjects diagnosed with spastic diplegic cerebral palsy and crouch gait will be recruited and ten healthy controls will be recruited in this study with inform consents. Detailed physical examination and motion analysis experiments will be performed in normal group and in spastic diplegic patients before the hamstring lengthening and follow ip after six months. The subjects would be asked to perform level walking with self-selected pace and sit-to-stand from an armless chair. For each test, subjects would repeat at least 5 times, with their kinematic, kinetic and EMG data collected simultaneously. With thorough analysis and comparison of these data, it is hoped that a reference in clinical decision of hamstring lengthening can be established, and a complete knowledge of the effects after hamstring lengthening, which will be helpful for future clinical rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* cerebral palsy
* couch gait

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2004-08; Study Completion 2005-07

PRIMARY OUTCOMES:
Gait
Sit-to-stand

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Ming Wang, MD, Study Chair — Dept. of Orthopaedic, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospitial, Taipei, Taiwan